CLINICAL TRIAL: NCT00906490
Title: Observational Clinical Study of the Intravenous Blood Glucose System in Hospitalized Adult Elective or Non-Emergent Surgery and Medical/Surgical Intensive Care Unit Patients
Brief Title: Clinical Study of the Intravenous Blood Glucose System in Hospitalized Adult Elective or Non-Emergent Surgery and Medical/Surgical Intensive Care Unit Patients
Status: Completed | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Collaborators: DexCom, Inc. (Industry); Medical Device Consultants, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2008-11
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Last update posted 2013-08-20 (Estimated); Status verified 2013-08

CONDITIONS: Blood Glucose
Keywords: Glucose Monitoring; Accurate Blood Glucose Monitoring in critical care setting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Intravenous Blood Glucose monitoring system — Insertion of blood glucose monitoring sensor into peripheral vascular IV line.

SUMMARY:
The primary objective of this study is to evaluate the performance and safety of the intravenous blood glucose (IVBG) System relative to point of care (POC) meter performance when each method is compared to the Yellow Springs Instrument (YSI) under various conditions in the operating room (OR), ICU and general ward (GW) in subjects undergoing elective or non-emergent surgery as well as subjects admitted to the medical/surgical ICU. POC meter systems are currently used in the hospital environment to measure blood glucose values. The YSI is an accepted reference standard for assessing POC meter accuracy.

The secondary objective of this study is to evaluate the performance of the IVBG System as compared with the YSI under various conditions in the operating room (OR), intensive care unit (ICU) and general ward (GW) in subjects undergoing elective or non-emergent surgery as well as subjects admitted to the medical/surgical ICU.

DETAILED DESCRIPTION:
Subjects will have their glucose values collected from the IVBG System and compared with paired plasma glucose measurements obtained using theYSI with comparative blood samples collected from a CVC, an arterial line or a peripheral vein.

* Blood samples collected per time point: approximately 2ml for waste and1mL for glucose measurement. In the event that a closed blood drawing system is utilized, the waste would be reduced or eliminated.
* The comparative blood samples will be drawn manually at a maximum frequency of once every four hours.
* Sample draws not to exceed 23 per subject for the duration of the study. This includes 18 comparative blood samples and 5 calibration samples to be draw as needed (e.g. recalibration). Including the partial thromboplastin time (PTT) draws described in section 3.1.2, there would be approximately 100 mL or 6.8 tablespoons drawn per subject. In the case where a closed blood drawing system is used consistently, this would be approximately 50 mL or 3.4 tablespoons per subject.

POC meter blood glucose measurements will be performed at the same time as the blood sample draws described above.

ELIGIBILITY:
Inclusion Criteria:

* ICU ≥ 24 hours
* sign ICF

Exclusion Criteria:

* transplant Pt
* brain injury/surgery
* DKA
* end stage disease
* restricted venous access
* hx of HITT
* contraindication for anti-coagulation Tx
* positive pregnancy test
* in other drug, device, or biologic study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute care facility patient with a minimum of 24 hour ICU stay.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
A non-inferior design to demonstrate that the IVBG System is equivalent (non-inferior) to a POC meter with respect to the proportion of glucose measurements that are deemed acceptable using a metric defined in ISO 15197. | During 72 hours of anticipated Sensor dwell time

SECONDARY OUTCOMES:
Accuracy of Device against YSI (Blood Glucose Analyser) | During 72 hours of anticipated Sensor dwell time

CONTACTS AND LOCATIONS:
Overall Officials: Grand Bochicchio, MD, Principal Investigator — University of Maryland Medical School
Locations (5):
- United States (5):
  - Washington Hospital Center (WHC), Washington D.C., District of Columbia
  - University of Maryland School of Medicine, Baltimore, Maryland
  - International Diabetes Center (IDC), Methodist Hospital, Minneapolis, Minnesota
  - Providence Heart and Vascular Institute, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania